CLINICAL TRIAL: NCT02368652
Title: A Randomized, Double-blind, Multi-center, Phase III Clinical Trial to Evaluate the Antihypertensive Efficacy and Safety of Amlodipine Besylate and Candesartan Cilexetil Combination in Patients With Essential Hypertension Who Are Not Adequately Controlled With Candesartan Cilexetil Monotherapy
Brief Title: A Study to Evaluate the Efficacy and Safety of Amlodipine Besylate and Candesartan Cilexetil in Essential Hypertension Patient Who Are Not Adequately Controlled With Candesartan Cilexetil Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_CCA_301A
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CC 16mg (Experimental): Candesartan ceilexetil 16mg, once a day for 8 weeks
  Interventions: Drug: Candesartan cilexetil 16mg
- AML 10mg / CC 16mg (Experimental): Amlodipine 10mg and Candesartan ceilexetil 16mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 10mg, Candesartan cilexetil 16mg

INTERVENTIONS:
Drug: Candesartan cilexetil 16mg — Daily oral administration for 8 weeks
  Other Names: Atacand 16mg
  Arms: CC 16mg
Drug: Amlodipine 10mg, Candesartan cilexetil 16mg — Daily oral administration for 8 weeks
  Other Names: Norvasc 10mg, Atacand 16mg
  Arms: AML 10mg / CC 16mg

SUMMARY:
Compare the safety and efficacy of amlodipine besylate and candesartan cilexetil combination therapy on patients of essential hypertension who are not properly controlled by candesartan cilexetil monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 19 and ≤ 75 years old
* Subject with essential hypertension
* Subject who have voluntarily agreed to participate in the trial and signed the written informed consent form, after having listened to the purpose, method, and effect of the clinical trial

Exclusion Criteria:

* Subject who is siDBP ≥ 120 mmHg or siSBP ≥ 200 mmHg at Visit 1 (screening)
* Subject with difference in the mean blood pressure of over 10 mmHg for siDBP or 20 mmHg for siSBP between both arms at the screening visit
* Subject with known or suspected secondary hypertension [Including but not limited to any of the following: renovascular diseases, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, primary hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromo-cytoma, polycystic kidney disease, etc.]
* Subject with symptomatic orthostatic hypotension(a sudden fall in siDBP of at least 10 mmHg or siSBP of at least 20 mmHg after standing compared with blood pressure from the sitting or supin position)
* Subject with type 1 or type 2 diabetes mellitus with poor glucose control (defined as subject on inculin treatment, with HbA1c > 9.0% or with a modification in the oral anti-hyperglycemic medication regiment within the past 12 weeks prior to visit 1)
* Subject with severe heart disease(congestive heart failure(NYHA class 3 or 4), ischemic heart disease within the past 6 months(unstable angina, myocardial infarction), peripheral blood vascula disease, history of Percutaneous Transluminal Coronary Angioplasty or coronary artery bypass grafting)
* Subject with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically significant arrhythmia
* Subject with hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, haemodynamically relevant stenosis of the aortic or mitral valve
* Subject with cardiogenic shock
* Subject with severe cerebrovascular disease (history of stroke, cerebral infraction, or cerebral hemorrhage within the past 6 months)
* Subject with a history of or ongoing wasting disease, autoimmune diseases(rheumatoid arthritis, systemic lupus erythematosus, etc.) or connective tissue disease
* Subject with known moderate or malignant retinopathy (history of retinal signs of hemorrhage, visual impairment, retinal microaneurysm etc. within the past 6 months)
* Subject with any surgical or medical condition of the gastrointestinal tract that might sugnificantly alter the absorption, distribution, metabolism or excretion of the drug
* Subject with a history of malignant tumors including leukemia and lymphoma within the past 5 yesrs(except for localized basal cell carcinoma of the skin)
* Subject with any chronic inflammatory condition needing chronic anti-inflammatory therapy
* Subject with chronic kidney disase on dialysis
* Subject with the following clinically significant laboratory abnormalities:

  * AST or ALT > 3 x Upper Limit Normal(ULN)
  * Serum Creatinine > 1.5 ULN
  * Serum potassium < 3.5 mmol/L or > 5.5mmol/L
* Subject requiring concomitant use of other antihypertensive or contraindicated drugs during the entire study period
* Subject with known or suspected contraindications, including history of allergy or hypersensitivity to ARB or dihydropyridine derivatives
* Subject who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or ARB
* Pregnant women or lactating mother, women suspected of being pregnant, women who wish to be pregnant during the study or women of child-bearing potential who are not using medically acceptable methods of contraception (oral contraceptinve, intra-uterine device, condom, etc.), except for women with surgical sterilization. Pre-menopausal women who are not surgically sterilized must have a negative pregnancy test result at Visit1 and maintain acceptable methods of contraception throughout the study. preiodic abstinence (eg. symptothermal, calendar, post-ovulation methods), or hormonal contraceptive are not acceptable methods of contraception
* History of drug or alcohol abuse within the past 1 year
* Use of other investigational products within the past 4 weeks
* Subject who are jdged unsuitable to participate in the study in the opinion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in sitting Diastolic Blood Pressure (siDBP) at week 8 compared to baseline | Week 8

SECONDARY OUTCOMES:
Change in siDBP at week 4 | Week 4
Change in sitting Systolic Blood Pressure (siSBP) at week 4 and 8 | Week 4 and 8
Proportion of patients achieving ΔsiDBP ≥ 10 mmHg and ΔsiSBP ≥ 20 mmHg after 8 weeks | Week 8
Proportion of patients achieving siDBP < 90 mmHg and siSBP < 140 mmHg after 8 weeks | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Seungjae Tahk, Principal Investigator — Ajou University School of Medicine
Locations (19):
- South Korea (19):
  - Hallym University Sungsim Hospital, Anyang-si
  - Inje University Busan Baik Hospital, Busan
  - Inje University Haeundae Baik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Baik Hospital, Ilsan
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Gangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul Medical Center, Seoul
  - Seoul St. Mary's Hospital Catholic University, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju